CLINICAL TRIAL: NCT00000471
Title: Lifestyle Heart Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 60; R01HL042554 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2000-01

CONDITIONS: Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases; Hypercholesterolemia; Hypertension; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Heart Diseases; Hypercholesterolemia; Hypertension; Myocardial Ischemia | interventions — Diet; Diet, Vegetarian; Diet, Fat-Restricted; Exercise

INTERVENTIONS:
Behavioral: diet, vegetarianism
Behavioral: diet, fat-restricted
Behavioral: exercise
Behavioral: smoking cessation

SUMMARY:
To assess long-term effects of a strict lifestyle change program on lipids, blood pressure, myocardial perfusion, and coronary atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

The trial was the first randomized, controlled trial to determine whether patients outside a hospital could be motivated to make and sustain comprehensive lifestyle changes and whether coronary disease regression could occur as a result of lifestyle changes alone.

DESIGN NARRATIVE:

Patients were randomly assigned to an experimental group or to a usual-care group. Experimental-group patients were prescribed a lifestyle program including a low-fat vegetarian diet, moderate aerobic exercise, stress management training, stopping smoking, and group support. No animal products were allowed in the vegetarian diet except egg white and one cup per day of non-fat milk or yogurt. The diet contained approximately 10 percent of calories as fat. Control-group patients were not asked to make lifestyle changes. Coronary angiography was performed at baseline and at one year to assess progression or regression of disease. Patients were recruited into the trial between January 1986 and November 1988. The trial was supported prior to April 1989 from various sources other than the National Heart, Lung, and Blood Institute. Follow-up continued for four years.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
Men and women, ages 35 to 75, with angiographically documented one, two, or three vessel coronary disease; no myocardial infarction during the preceeding six weeks; and not receiving streptokinase, alteplase, or lipid-lowering drugs.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1989-04; Study Completion 1993-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Gould — University of Texas; Dean Ornish — University of California School of Medicine

REFERENCES:
- [Background] Ornish D, Brown SE, Scherwitz LW, Billings JH, Armstrong WT, Ports TA, McLanahan SM, Kirkeeide RL, Brand RJ, Gould KL. Can lifestyle changes reverse coronary heart disease? The Lifestyle Heart Trial. Lancet. 1990 Jul 21;336(8708):129-33. doi: 10.1016/0140-6736(90)91656-u. PMID 1973470
- [Background] Gould KL, Ornish D, Kirkeeide R, Brown S, Stuart Y, Buchi M, Billings J, Armstrong W, Ports T, Scherwitz L. Improved stenosis geometry by quantitative coronary arteriography after vigorous risk factor modification. Am J Cardiol. 1992 Apr 1;69(9):845-53. doi: 10.1016/0002-9149(92)90781-s. PMID 1550011
- [Background] Gould KL, Ornish D, Scherwitz L, Brown S, Edens RP, Hess MJ, Mullani N, Bolomey L, Dobbs F, Armstrong WT, et al. Changes in myocardial perfusion abnormalities by positron emission tomography after long-term, intense risk factor modification. JAMA. 1995 Sep 20;274(11):894-901. doi: 10.1001/jama.1995.03530110056036. PMID 7674504